CLINICAL TRIAL: NCT05302869
Title: Perceptions of Physiotherapy and Rehabilitation Department Students and Graduated Physiotherapists About Their Professions
Brief Title: Perceptions of Physiotherapy and Rehabilitation Professions
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Nuray Alaca, Assoc Prof. Nuray Alaca, Acibadem University
Other Study IDs: ATADEK-2022-01-11
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Perception, Self; Physiotherapy
Keywords: Perception, Self; Physiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Students
  Interventions: Other: None intervention
- Physiotherapist
  Interventions: Other: None intervention

INTERVENTIONS:
Other: None intervention — None intervention

SUMMARY:
In this study, it is aimed to determine the perspectives and satisfaction of the students of the Physiotherapy and Rehabilitation Department about the physiotherapist profession, and to compare these results according to the class periods.

Our secondary aim is to determine the perspectives and satisfaction of graduate physiotherapists towards the physiotherapist profession and to compare these results according to their graduation years.

ELIGIBILITY:
Inclusion Criteria:

* Students in the physiotherapy and rehabilitation department or become a graduate physiotherapist

Exclusion Criteria:

* Students or a graduate physiotherapist with serious mental illness

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: The current study will be conducted by face-to-face interviews within the scope of questionnaires prepared by us for students Students or a graduate physiotherapist
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Perceptions of students/physiotherapist about the physiotherapist profession | Baseline time
  Measuring perceptions of physiotherapist and other professions relative to each other (0-10). low scores indicate poor perception, high scores indicate good perception. [the minimum (8 point) and maximum values (80 point)], higher scores were mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nuray ALACA, Principal Investigator — Acibadem University
Locations (1):
- Acibadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided